CLINICAL TRIAL: NCT02590926
Title: Safety of Negative FrActional Flow Reserve in Patients With ChallEnging Lesions
Acronym: FACE
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Claudio Moretti, Head, Cardiology Cath Lab, A.O.U. Città della Salute e della Scienza
Other Study IDs: 370/2015
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Fractional Flow Reserve, Myocardial
Keywords: Fractional Flow Reserve, Myocardial
MeSH Terms: interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients: patients with stable angina and/or documented ischemia presenting with:
  * An angiographic stenosis of more than 50% and less than 90% of the left main
  * Any proximal descending anterior with a stenosis of more than 50% and less than 90%
  * Two or three vessel disease with a stenosis of more than 50% and less than 90% and a left ventricle ejection fraction less than 40%
  * Single remaining patent coronary artery with stenosis >50% and less than 90%
  Interventions: Procedure: Fractional Flow Reserve, Myocardial

INTERVENTIONS:
Procedure: Fractional Flow Reserve, Myocardial — The ratio of maximum blood flow to the myocardium with coronary stenosis present, to the maximum equivalent blood flow without stenosis.

SUMMARY:
Fractional Flow Reserve (FFR) has recently emerged and has been largely validated as a safe and efficacious way of ischemia testing for patients with stable angina. The new recently ESC guidelines have strongly suggested a FFR based approach for patients with stable angina, also for those with challenging lesions like left main disease, severe multivessel stenosis for heart failure patients and those with single remaining vessels although left main disease and an ejection fraction less than 30% are exclusion criteria of the randomized controlled trials on this topic. Consequently the investigators performed a prospective multicenter study to understand the safety and efficacy of a FFR based approach for these patients.

DETAILED DESCRIPTION:
The present is a multicenter prospective study enrolling all patients with stable angina and/or documented ischemia presenting with:

* An angiographic stenosis of more than 50% and less than 90% of the left main
* Any proximal descending anterior with a stenosis of more than 50% and less than 90%
* Two or three vessel disease with a stenosis of more than 50% and less than 90% and a left ventricle ejection fraction less than 40%
* Single remaining patent coronary artery with stenosis >50% and less than 90%

In all of these patients FFR (Fractional Flow Reserve) will be performed according to guidelines and stenting will be performed or deferred according to the result of this test. Other techniques, like iFR, IVUS and OCT will be left at the operators' choice and will be recorded. MACE (a composite end point of death, myocardial infarction and target vessel revascularization and stent thrombosis) will be the primary end point, while its single components will be the secondary ones.

ELIGIBILITY:
Inclusion Criteria:

* An angiographic stenosis of more than 50% and less than 90% of the left main
* Any proximal descending anterior with a stenosis of more than 50% and less than 90%
* Two or three vessel disease with a stenosis of more than 50% and less than 90% and a left ventricle ejection fraction less than 40%
* Single remaining patent coronary artery with stenosis >50% and less than 90%

Exclusion Criteria:

* Severe aortic stenosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with stable angina
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2014-09-26; Primary Completion 2016-09-05 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
MACE | 3 years
  composite end point of death, myocardial infarctio, target vessel revascularization and target lesion revascularization, stent thrombosis
TVF (only for deferred lesion) | 1 and 2 years
  composite of cardiac death,myocardial infarction and target vessel revascularization due to deferred lesion

SECONDARY OUTCOMES:
Death | 1 and 2 years
  and also cardiac death as a separate outcome
TLR | 1 and 2 years
AMI | 1 and 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fabrizio D'Ascenzo, Turin, Italy

REFERENCES:
- [Result] Layland J, Oldroyd KG, Curzen N, Sood A, Balachandran K, Das R, Junejo S, Ahmed N, Lee MM, Shaukat A, O'Donnell A, Nam J, Briggs A, Henderson R, McConnachie A, Berry C; FAMOUS-NSTEMI investigators. Fractional flow reserve vs. angiography in guiding management to optimize outcomes in non-ST-segment elevation myocardial infarction: the British Heart Foundation FAMOUS-NSTEMI randomized trial. Eur Heart J. 2015 Jan 7;36(2):100-11. doi: 10.1093/eurheartj/ehu338. Epub 2014 Sep 1. PMID 25179764
- [Result] De Bruyne B, Fearon WF, Pijls NH, Barbato E, Tonino P, Piroth Z, Jagic N, Mobius-Winckler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd K, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Limacher A, Nuesch E, Juni P; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI for stable coronary artery disease. N Engl J Med. 2014 Sep 25;371(13):1208-17. doi: 10.1056/NEJMoa1408758. Epub 2014 Sep 1. PMID 25176289
- [Result] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Result] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Derived] Barbero U, D'Ascenzo F, Campo G, Kleczynski P, Dziewierz A, Menozzi M, Jimenez Diaz VA, Cerrato E, Raposeiras-Roubin S, Ielasi A, Rognoni A, Fineschi M, Kanji R, Jaguszewski MJ, Picchi A, Ando G, Soraci E, Mancone M, Sardella G, Calcagno S, Gallo F, Huczek Z, Krakowian M, Verardi R, Montefusco A, Omede P, Lococo M, Moretti C, D'Amico M, Rigattieri S, Gaita F, Rinaldi M, Escaned J. Safety of FFR-guided revascularisation deferral in Anatomically prognostiC diseasE (FACE: CARDIOGROUP V STUDY): A prospective multicentre study. Int J Cardiol. 2018 Nov 1;270:107-112. doi: 10.1016/j.ijcard.2018.06.013. Epub 2018 Jun 8. PMID 29937300